CLINICAL TRIAL: NCT01454024
Title: A Study Evaluating the Safety of NovoPen®3 and FlexPen® in Subjects With Type 1 and Type 2 Diabetes. A 24-week, Prospective, Multi-centre, Open-labelled, Non-interventional Study
Brief Title: Evaluating Safety of NovoPen® 3 and/or FlexPen® Devices in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-3882; U1111-1116-2517 (Other: WHO)
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total study population
  Interventions: Device: FlexPen®; Device: NovoPen® 3

INTERVENTIONS:
Device: FlexPen® — Prescribed insulin treatment delivered by FlexPen® as part of routine clinical practice
Device: NovoPen® 3 — Prescribed insulin treatment delivered by NovoPen® 3 as part of routine clinical practice

SUMMARY:
This study is conducted in Asia. The aim of of this study is to evaluate the safety of NovoPen® 3 and/or FlexPen® devices (if available on the market) measured by the number of adverse events and technical complaints in patients with type 1 and type 2 diabetes in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Any subjects who are previously using Actrapid®, Insulatard®, and Mixtard® 30 with vial / NovoLet® or insulin human with ErgoPen®2 for type 1 and type 2 diabetes treatment, will be eligible for the study after the physician has taken the decision to use study insulin products with the study devices

Exclusion Criteria:

* Subjects treated with Actrapid® Penfill®, Insulatard® Penfill®, or Mixtard® 30 Penfill® with NovoPen®3 or Actrapid® FlexPen®, Insulatard® FlexPen®, or Mixtard® 30 FlexPen® for more than 4 weeks before inclusion into this study
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to insulin human or to any of the excipients
* Women who are pregnant, breast feeding or have the intention of becoming pregnant within the next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The selection of the subjects will be at the discretion of the individual physician based on clinical judgement.
Sampling Method: Non-Probability Sample
Enrollment: 1031 (Actual)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and technical complaints | Week 0-24

SECONDARY OUTCOMES:
Number of adverse drug reactions (ADR) including hypoglycaemic events | Week 0-12, week 24
Number of serious adverse drug reactions including major hypoglycaemic events | Week 0-12, week 24
HbA1c (haemoglobin A1c) | Week 0, week 12 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Karachi, Pakistan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com